CLINICAL TRIAL: NCT04715009
Title: The Effect of Smartphone Use on Neck Flexion Angle and Hand Grip Power Among Adolescence
Brief Title: Smartphone Use and Neck Flexion Angle
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Nehad Ahmed Youness Abo-zaid, lecturer ofphysical terapy, South Valley University
Other Study IDs: Smartphone
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Neck Disorder
Keywords: smartphone; neck flexion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- participants use smartphone less than 4 hours per day: participants use smartphone less than 4 hours per day
- participants use smartphone more than 4 hours per day: participants use smartphone more than 4 hours per day

SUMMARY:
Excessive smartphone use can disrupt your sleep, which can have a serious impact on your overall mental health. It can impact your memory, affect your ability to think clearly, and reduce your cognitive and learning skills. Encouraging self-absorption.

DETAILED DESCRIPTION:
Persistent failed attempts to use cell phone less often. Preoccupation with smartphone use. Turns to cell phone when experiencing unwanted feelings such as anxiety or depression. Excessive use characterized by loss of sense of time.

Nomophobia-an abbreviation of "no-mobile-phone-phobia"-is also called "cell phone addiction." Symptoms include: Experiencing anxiety or panic over losing your phone. Obsessively checking for missed calls, emails, and texts.

ELIGIBILITY:
Inclusion Criteria:

* volunteers using smartphone less or more than 4 hours per day

Exclusion Criteria:

* low back pain surgeries affecting upper limps

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: healthy volunteers using smartphone less or more than 4 hours per day have not any signes of musculoskeletal problems
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
the neck flexion angle | the neck flexion angle at day 0
  flexion angle of the neck
the neck flexion angle | the neck flexion angle at day 120
  flexion angle of the neck

SECONDARY OUTCOMES:
hand grip power | power of hand at date 0
  power of hand
hand grip power | power of hand at date 120
  power of hand

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A Abo-zaid, lecturer, Principal Investigator — South Valley University, Faculty of Physical Therapy
Locations (1):
- Nehad ahmed youness, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonney RA, Corlett EN. Head posture and loading of the cervical spine. Appl Ergon. 2002 Sep;33(5):415-7. doi: 10.1016/s0003-6870(02)00036-4. PMID 12236650
- [Background] Janwantanakul P, Sitthipornvorakul E, Paksaichol A. Risk factors for the onset of nonspecific low back pain in office workers: a systematic review of prospective cohort studies. J Manipulative Physiol Ther. 2012 Sep;35(7):568-77. doi: 10.1016/j.jmpt.2012.07.008. Epub 2012 Aug 24. PMID 22926018
- [Background] Hansraj KK. Assessment of stresses in the cervical spine caused by posture and position of the head. Surg Technol Int. 2014 Nov;25:277-9. PMID 25393825
- [Background] Grimmer-Somers K, Milanese S, Louw Q. Measurement of cervical posture in the sagittal plane. J Manipulative Physiol Ther. 2008 Sep;31(7):509-17. doi: 10.1016/j.jmpt.2008.08.005. PMID 18804001